CLINICAL TRIAL: NCT02328755
Title: Targeting Cross-presentation With Peginterferon Alfa-2a to Enhance Anti-leukemic Responses After Allogeneic Transplantation in High Risk Acute Myeloid Leukemia
Brief Title: Peginterferon Alfa-2a to Enhance Anti-leukemic Responses After Allogeneic Transplantation in Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2014.107; HUM00093471 (Other: University of Michigan)
Record Dates: First submitted 2014-11-11; First posted 2014-12-31 (Estimated); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — peginterferon alfa-2a; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- peg-IFN-α (Experimental): peg-IFN-α will be administered prior to HCT (Hematopoietic Cell Transplant) and at three subsequent time points post HCT. (Maximum of 4 doses) It will be administered by subcutaneous injection every 14 days beginning with dose level 1.
  Dose Level -1 - 45mcg Dose Level 1 - 90mcg Dose Level 2 - 180 mcg
  Interventions: Drug: peg-IFN-α; Procedure: Hematopoietic Cell Transplant (HCT); Drug: Tacrolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: peg-IFN-α
  Other Names: PEGASYS®
Procedure: Hematopoietic Cell Transplant (HCT)
Drug: Tacrolimus — Calcineurin inhibitor administered along with HCT for Graft Versus Host Disease (GVHD) prophylaxis. Cyclosporine may be substituted if patients cannot tolerate tacrolimus.
Drug: Methotrexate — Administered along with HCT for Graft Versus Host Disease (GVHD) prophylaxis.

SUMMARY:
This protocol is an open label, single arm, non-randomized, phase I / II clinical trial investigating the use of pegylated interferon alpha-2a (peg-IFN-α, Pegasys®, Genentech) for prevention of relapse in acute myeloid leukemia (AML) not in remission at the time of allogeneic hematopoietic stem cell transplantation (HCT).

DETAILED DESCRIPTION:
This protocol is an open label, single arm, non-randomized, phase I / II clinical trial investigating the use of pegylated interferon alpha-2a (peg-IFN-α, Pegasys®, Genentech) for prevention of relapse in acute myeloid leukemia (AML) not in remission at the time of allogeneic hematopoietic stem cell transplantation (HCT). The inability to attain remission status following induction therapy for AML remains a significant problem and is associated with poor outcomes. While HCT remains a curative option, its activity in the setting of relapsed or refractory AML is significantly diminished due to high relapse.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have AML not in remission or at very high risk for HCT (Hematopoietic Cell Transplantation) relapse.
* For newly diagnosed AML, patients must have achieved two consecutive induction attempts without achieving complete remission
* For patients initially in complete remission whose AML relapses > 6 months after preceding remission, one re-induction must be attempted to be eligible
* For AML patients with early relapse, in whom the preceding remission is shorter than 6 months duration, no re-induction regimen is necessary to be eligible
* Patients with antecedent MDS (Myelodysplastic Syndrome) who progress to AML may have therapies rendered during both phases counted towards these requirements.
* Patients with poor cytogenetic or molecular risk associated with very high risk for relapse after HCT may proceed without provisions for prior treatment. However, they must have received at least one induction attempt.
* Patients must be ≥ 18 years of age and considered a candidate for HCT
* Karnofsky ≥ 70% (Karnofsky performance status is measure of a cancer patients general well being and activities of daily life. Scores range from 100 to 0 where 100 is perfect health and 0 is death
* Patients must meet acceptable organ function criteria: Total Bilirubin ≤2.5 mg%; AST (Aspartate transaminase) and ALT (Alanine transaminase) <5.0 X institutional upper limit of normal; GFR (Glomerular filtration rate) >40 mL/min/1.73 m2 for patients with creatinine levels above institutional normal; Lung function tests (DLCO, FEV1, FVC) > 50%; Ejection fraction > 50%
* All patients must sign an informed consent
* Women and men of child-bearing potential must agree to use adequate contraception

Exclusion Criteria:

* Prior chemotherapy treatment for AML within 21 days from the initiation of HCT conditioning
* Patients may NOT have evidence or symptoms of CNS disease at the time of enrollment
* HIV or HTLV1 / HTLV2 (Human T-lymphotrophic virus) (seropositivity and/or PCR positivity)
* Patients less than 18 years of age
* Pregnant and nursing mothers are excluded from this study
* Patients with untreated or uncontrolled neuropsychiatric illness
* Any physical or psychological condition that, in the opinion of the investigator, would pose unacceptable risk to the patient
* Uncontrolled infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-01; Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Magenau, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Magenau JM, Peltier D, Riwes M, Pawarode A, Parkin B, Braun T, Anand S, Ghosh M, Maciejewski J, Yanik G, Choi SW, Talpaz M, Reddy P. Type 1 interferon to prevent leukemia relapse after allogeneic transplantation. Blood Adv. 2021 Dec 14;5(23):5047-5056. doi: 10.1182/bloodadvances.2021004908. PMID 34607341

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One person did not start study treatment; no participants were assigned or de-escalated to Dose Level -1 (45mcg).
Groups:
- Dose Level 1, 90 mcg Peg-IFN-α: 90 mcg peg-IFN-α administered prior to hematopoietic cell transplantation (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days.
- Dose Level 2, 180 mcg Peg-IFN-α: 180 mcg peg-IFN-α administered prior to hematopoietic cell transplantation (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days.
Period: Overall Study
Arm/Group | Dose Level 1, 90 mcg Peg-IFN-α | Dose Level 2, 180 mcg Peg-IFN-α
Started | 3 | 33
Completed (Evaluable for the phase II primary endpoint of relapse at 6-months post-HCT) | 0 (Evaluable for the phase II primary endpoint of relapse at 6-months post-HCT) | 31
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1 - 90 mcg Peg-IFN-α: Dose Level 1 - 90 mcg peg-IFN-α administered prior to hematopoietic cell transplant (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days beginning with dose level 1.
- Dose Level 2 - 180 mcg Peg-IFN-α: Dose Level 2 - 180 mcg peg-IFN-α administered prior to hematopoietic cell transplant (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days beginning with dose level 1.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - 90 mcg Peg-IFN-α | Dose Level 2 - 180 mcg Peg-IFN-α | Total
Number analyzed (Participants) | 3 | 33 | 36
Age, Continuous [Median (Full Range); unit: years] | 56 [54 to 67] | 60 [17 to 72] | 60 [17 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 13 | 14
  Male | 2 | 20 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 33 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 32 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 33 | 36
Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI)CT-Cl [Median (Full Range); unit: units on a scale] — The HCT-CI is a comorbidity index that comprises 17 different categories of organ dysfunction. Positive findings are summed into a total score, ranging from 0 to 29, where 0 is no comorbidity or concern, and higher numbers indicate serious related concerns, with 3 or more being high risk.
  units on a scale | 5 [4 to 5] | 3 [0 to 7] | 3 [0 to 7]
Disease Status at HCT [Count of Participants; unit: Participants]
  Not in remission | 3 | 32 | 35
  Remission | 0 | 1 | 1
Cytogenic risk [Count of Participants; unit: Participants]
  Poor | 2 | 16 | 18
  Intermediate | 1 | 16 | 17
  Unknown | 0 | 1 | 1
Disease Risk Score [Count of Participants; unit: Participants] — as per Duval et al. J. Clin. Oncol 2010; 28(23): 3730-8. This scale is designed to predict the overall survival. The score is on a range from 0 to 6, where 0 is no risk and 6 is highest.
  Participants
    Greater or equal to 3 | 2 | 19 | 21
    2 | 1 | 11 | 12
    1 | 0 | 3 | 3
Time to HCT from AML Diagnosis [Median (Full Range); unit: days] | 98 [55 to 2051] | 192 [61 to 1996] | 142 [55 to 2051]
Donor Type [Count of Participants; unit: Participants]
  Unrelated | 2 | 18 | 20
  Related | 1 | 15 | 16
Human Leukocyte Antigen match [Count of Participants; unit: Participants]
  Yes | 3 | 31 | 34
  No | 0 | 2 | 2
Donor Source [Count of Participants; unit: Participants]
  Peripheral Blood Stem Cells | 2 | 29 | 31
  Bone Marrow | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Peg-IFN-α
Description: The dose level assigned to the most participants is selected as the MTD. Participants from the arms for dose level 1 (90mcg, 3 participants) and dose level 2 (180mcg, 33 participants) were analyzed together to determine the MTD. Dosage levels are determined by dose-limiting toxicities (DLTs). Only DLTs encountered during the treatment period, prior to day 56 post HCT (or 14 days after final treatment, whichever comes later), are counted. DLTs after the treatment period are counted only if they reflect an ongoing toxicity that initiated in the treatment period.
Time Frame: Up to day 56 post-transplant or up to 14 days after final treatment with peg-IFN-α, whichever comes later. Data was collected up to 63 days.
Population: All participants (n=36)
Measure: Number; unit: mcg
Groups:
- Peg-IFN-α: peg-IFN-α was administered prior to HCT (Hematopoietic Cell Transplant) and at three subsequent time points post HCT. (Maximum of 4 doses) It was administered by subcutaneous injection every 14 days beginning with dose level 1.
  Dose Level -1 - 45mcg Dose Level 1 - 90mcg Dose Level 2 - 180 mcg peg-IFN-α It was begun at 90 mcg, would have been reduced back to 45 mcg if necessary, and after 3 participants it was increased to 180 mcg.
Arm/Group | Peg-IFN-α
Number analyzed (Participants) | 36
mcg | 180

2. Primary Outcome: Phase 2: Number of Patients That Relapse
Description: The cumulative incidence of relapse, estimated using proportional hazard model for the competing risk of non-relapse mortality (NRM).
Time Frame: 6 Months Post HCT
Population: The first row shows analysis for recipients of HLA-matched HCT who received the phase II MTD (180mcg) peg-IFN-α (n=31); the second row shows all participants (n=36)
Measure: Number; unit: percentage of participants
Groups:
- Dose Level 1 - 90 mg Peg-IFN-α: 90 mcg peg-IFN-α administered prior to hematopoietic cell transplantation (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days.
- Dose Level 2 - 180 mg Peg-IFN-α: 180 mcg peg-IFN-α administered prior to hematopoietic cell transplantation (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days.
Arm/Group | Dose Level 1 - 90 mg Peg-IFN-α | Dose Level 2 - 180 mg Peg-IFN-α
Number analyzed (Participants) | 3 | 33
percentage of participants
  Phase II MTD (180mcg) participants with fully matched donor HCT: number analyzed (Participants) | 0 | 31
  Phase II MTD (180mcg) participants with fully matched donor HCT |  | 39
  All participants | 67 | 39
Statistical Analysis 1: Comparison: Dose Level 2 - 180 mg Peg-IFN-α; The analysis applies only to the first row, for recipients of HLA-matched HCT who received the phase II MTD (180mcg) peg-IFN-a (n=31); Test type: Other — Single group; cumulative incidence = 0.39, 95% CI 2-sided [0.24 to 0.58]

3. Secondary Outcome: Phase 2: Overall Survival Time
Description: Estimated using Kaplan-Meier methods, overall survival (OS) will be calculated from the day of transplantation (day 0) until death; shown at 6 month and 2 year estimates
Time Frame: 1 year or until study stops, whichever is later. Median time of follow-up was 25 months.
Population: Some rows show analysis for recipients of HLA-matched HCT who received the phase II MTD (180mcg) peg-IFN-α(n=31); for 6 month data, the additional row shows all participants (n=36)
Measure: Number; unit: percentage of participants
Groups:
- Dose Level 1 - 90 mcg Peg-IFN-α: 90 mcg peg-IFN-α administered prior to hematopoietic cell transplantation (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days.
- Dose Level 2 - 180 mcg Peg-IFN-α: 180 mcg peg-IFN-α administered prior to hematopoietic cell transplantation (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days.
Arm/Group | Dose Level 1 - 90 mcg Peg-IFN-α | Dose Level 2 - 180 mcg Peg-IFN-α
Number analyzed (Participants) | 3 | 33
percentage of participants
  6 months (Phase II MTD [180 mcg] participants with fully matched donor HCT): number analyzed (Participants) | 0 | 31
  6 months (Phase II MTD [180 mcg] participants with fully matched donor HCT) |  | 55
  6 months - all participants | 33 | 55
  2 years (Phase II MTD [180 mcg] participants with fully matched donor HCT): number analyzed (Participants) | 0 | 31
  2 years (Phase II MTD [180 mcg] participants with fully matched donor HCT) |  | 33
Statistical Analysis 1: Comparison: Dose Level 2 - 180 mcg Peg-IFN-α; The analysis applies only to the first row, data at 6 months, for recipients of HLA-matched HCT who received the phase II MTD (180mcg) peg-IFN-a (n=31); Test type: Other — Single group; Kaplan-Meier = 55, 95% CI 2-sided [40 to 75]; Survival proportion estimates at 6 months and 2 years were calculated using Kaplan-Meier methods, and the 2-sided, 95% confidence intervals calculated by the Greenwood method
Statistical Analysis 2: Comparison: Dose Level 2 - 180 mcg Peg-IFN-α; The analysis applies only to the 3rd row, data at 24 months, for recipients of HLA-matched HCT who received the phase II MTD (180mcg) peg-IFN-a (n=31); Test type: Other — Single group; Kaplan-Meier = 33, 95% CI 2-sided [19 to 58]; [other analysis details as in outcome 3, analysis 1]

4. Secondary Outcome: Phase 2: Event Free Survival Time
Description: Defined for this study as Leukemia Free Survival, and estimated using Kaplan-Meier methods.
Time Frame: 1 year or until study stops, whichever is later. Median time of follow-up was 25 months.
Population: Recipients of HLA-matched HCT who received phase II MTD (180mcg) peg-IFN-α (n=31)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Peg-IFN-α: peg-IFN-α was administered prior to HCT (Hematopoietic Cell Transplant) and at three subsequent time points post HCT. (Maximum of 4 doses) It was administered by subcutaneous injection every 14 days beginning with dose level 1.
  Dose Level 1 - 90 mcg Dose Level 2 - 180 mcg peg-IFN-α
Arm/Group | Peg-IFN-α
Number analyzed (Participants) | 31
percentage of participants
  6 months | 48 [34 to 70]
  2 years | 28 [15 to 52]
Statistical Analysis 1: Comparison: Peg-IFN-α; Test type: Other — Single group; [other analysis details as in outcome 3, analysis 1]

5. Secondary Outcome: Acute GVHD
Description: Grade 2-4 Acute GVHD estimated using proportional hazards ratio. Graded according to CTCAE v. 4.0; higher grades represent more severe events.
Time Frame: 6 months
Population: Recipients of HLA-matched HCT who received phase II MTD (180mcg) peg-IFN-a (n=31)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 180mcg Peg-IFN-α, HLA-matched: 180 mcg peg-IFN-a administered prior to hematopoietic cell transplantation (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days
Arm/Group | 180mcg Peg-IFN-α, HLA-matched
Number analyzed (Participants) | 31
percentage of participants | 39 [24 to 58]
Statistical Analysis 1: Comparison: 180mcg Peg-IFN-α, HLA-matched; Test type: Other — Single group; GVHD proportion estimates and corresponding 95% confidence intervals were calculated using methods of Fine and Gray

6. Secondary Outcome: Non-Relapse Mortality
Description: The cumulative incidence of non-relapse mortality is estimated by proportional hazard models methods.
Time Frame: 1 year or until study stops, whichever is later. Median time of follow-up was 25 months.
Population: Recipients of HLA-matched HCT who received phase II MTD (180mcg) peg-IFN-α (n=31)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 189mcg Peg-IFN-α, HLA-matched: 180 mcg peg-IFN-a administered prior to hematopoietic cell transplantation (HCT) and at three subsequent time points post HCT (maximum of 4 doses) every 14 days
Arm/Group | 189mcg Peg-IFN-α, HLA-matched
Number analyzed (Participants) | 31
percentage of participants
  6 months | 13 [5 to 31]
  2 years | 25 [12 to 46]
Statistical Analysis 1: Comparison: 189mcg Peg-IFN-α, HLA-matched; Test type: Other — Single group; Non-relapse mortality estimates and corresponding 95% confidence intervals were calculated using methods of Fine and Gray

ADVERSE EVENTS:
Time Frame: The assessment and reporting period for all adverse events will occur from the first day the treatment with peg-IFN-α is administered until day +56 post transplant or until 14 days after the last dose of peg-IFN-α is administered, whichever comes last. Adverse event data were collected up to 63 days. All-Cause Mortality assessed up to 4 years; median of 25 months.
Description: Only grade >=3 events were recorded; infectious disease and hematologic events were not included.
Groups:
- Phase I/Dose Level 1 - 90 mcg: peg-IFN-α 90 mcg administered prior to hematopoietic cell transplant (HCT) and at three subsequent time points post HCT (maximum of 4 doses), every 14 days. Tacrolimus: Calcineurin inhibitor administered along with HCT for Graft Versus Host Disease (GVHD) prophylaxis. Cyclosporine could be substituted if patients cannot tolerate tacrolimus. Methotrexate: Administered along with HCT for Graft Versus Host Disease (GVHD) prophylaxis.
- Phase 2/Dose Level 2 - 180 mcg Peg-IFN-α: peg-IFN-α 180 mcg administered prior to hematopoietic cell transplant (HCT) and at three subsequent time points post HCT (maximum of 4 doses), every 14 days. Tacrolimus: Calcineurin inhibitor administered along with HCT for Graft Versus Host Disease (GVHD) prophylaxis. Cyclosporine could be substituted if patients cannot tolerate tacrolimus. Methotrexate: Administered along with HCT for Graft Versus Host Disease (GVHD) prophylaxis.
Arm/Group | Phase I/Dose Level 1 - 90 mcg | Phase 2/Dose Level 2 - 180 mcg Peg-IFN-α
All-Cause Mortality (participants affected / at risk) | 2/3 | 22/33
Serious Adverse Events (participants affected / at risk) | 2/3 | 8/33
Other Adverse Events (participants affected / at risk) | 0/3 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I/Dose Level 1 - 90 mcg (N=3) | Phase 2/Dose Level 2 - 180 mcg Peg-IFN-α (N=33)
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Pneumonitis (ARDS) (1); Acute Hypoxemia (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 — consistent with gouty arthritis
Hypertension (Cardiac disorders) | 1 | 0
Hypotension (Cardiac disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Liver Function Test elevation (Hepatobiliary disorders) | 0 | 1
Graft Failure (Immune system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT02328755/Prot_SAP_000.pdf